CLINICAL TRIAL: NCT01971944
Title: The Influence of Beta Blocker Therapy on the Hemodynamic Response to Inotrope Infusion in Patients With Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1985
Record Dates: First submitted 2013-10-18; First posted 2013-10-30 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Acute Decompensated Heart Failure; Heart Failure
Keywords: Beta Blocker; Inotrope
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients achieving steady state concentrations of carvedilol: Patients achieving steady state concentrations of carvedilol who receive a trial of dobutamine followed by milrinone.
- Patients achieving steady state concentrations of metoprolol: Patients achieving steady state concentrations of metoprolol who receive a trial of dobutamine followed by milrinone.
- Patients not receiving beta blocker: Patients not receiving beta blocker who receive a trial of dobutamine followed by milrinone.

SUMMARY:
Purpose: To compare the hemodynamic effects of dobutamine and milrinone in hospitalized patients who are receiving Beta Blocker Participants: Patients who are admitted to the General Cardiology and Heart Failure Services at the University of North Carolina Hospitals with acute decompensated heart failure, who have maintained steady state concentrations of beta blocker therapy (carvedilol or metoprolol), and who are deemed by the health care team to require pulmonary artery catheter placement and inotropic therapy with dobutamine or milrinone by continuous infusion. Patients that are not currently receiving beta blocker therapy will be enrolled for comparative purposes; however, any patient not at steady state (on or off beta blocker therapy) will not be enrolled.

Procedures: After obtaining informed consent, patients will be assigned to the appropriate sub-study group based on beta blocker use (Study A: patients on stable doses of metoprolol and Study B: patients on stable doses of carvedilol). All patients should receive dobutamine followed by milrinone as outlined in the dosing algorithm (see inotrope dosing algorithm attached, as part of the usual standard of practice). Baseline pulmonary artery catheter hemodynamic parameters will be collected prior to administration of inotrope trial of dobutamine followed by milrinone. Hemodynamic parameters will be recorded per the dosing algorithm following initiation and dose titration. Dose titration will be determined by the health care team based upon patient response or lack thereof and tolerability. Changes in hemodynamic parameters in response to dobutamine or milrinone will be compared within study groups. Additionally, data will continue to be collected on patients receiving not beta blocker therapy for comparative purpose.

DETAILED DESCRIPTION:
Background:

First-line management of chronic heart failure includes beta blockers and angiotensin converting enzyme (ACE) inhibitors, as these agents have been shown to have significant benefits on morbidity and mortality in large clinical trials. Therefore, a substantial number of patients with chronic heart failure are receiving chronic beta blocker therapy, most commonly metoprolol succinate and carvedilol. However, despite significant advancements in the treatment of chronic heart failure, the natural history of the disease remains progressive and many patients develop acute decompensations requiring hospitalization. In the setting of acute decompensated heart failure, the use of inotropic agents may be required for hemodynamic support. The two most widely used inotropes are dobutamine and milrinone. Dobutamine primarily acts as a beta-1 receptor agonist with some effects on beta-2 and alpha-1 receptors. Milrinone is a phosphodiesterase III inhibitor, thus inhibiting the breakdown of cyclic adenosine monophosphate. As such, milrinone works at a site that is distal to beta receptors and may be less influenced by chronic beta blocker therapy. As such, one may speculate that the presence of a beta blocker would influence the hemodynamic response to dobutamine, but to a much lesser extent to milrinone, if at all.

Two small studies have assessed the hemodynamic response to dobutamine in the presence and absence of beta blocker therapy in patients with chronic heart failure. In addition, one of these studies assessed the response to enoximone, another phosphodiesterase III inhibitor. Both studies demonstrated that metoprolol did not significantly affect the hemodynamic response to dobutamine infusion, including its effect on cardiac index, heart rate, stroke volume, and systemic vascular resistance. Conversely, carvedilol was shown to have significant inhibitory effects on cardiac index, heart rate, and stroke volume during dobutamine infusion. In addition, carvedilol appeared to increase mean arterial pressure at higher doses of dobutamine. In the setting of an enoximone infusion, metoprolol increased the cardiac index and stroke volume responses, while maintaining other hemodynamic parameters. There was no significant difference in the hemodynamic response to enoximone infusion in the presence of carvedilol.

Why This Study is Needed:

Published studies that assessed the hemodynamic response to inotropes in the presence and absence of beta blockers included less than 50 patients combined. As such, the replication of their results is warranted in order to use this data to drive changes in clinical practice. Additionally, and equally as important, no study has been published, to the best of our knowledge, which has assessed the hemodynamic response to milrinone in the presence of metoprolol. . Although enoximone is a phosphodiesterase III inhibitor and is theoretically similar to milrinone, it is not approved for use in the United States, thus making it difficult to extrapolate these findings to milrinone. Lastly, the severity of illness in patients included in current literature does not reflect individuals who will receive the most benefit from therapy i.e. patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age and English-speaking who are admitted to the General Cardiology or Heart Failure Services at the University of North Carolina Hospitals with acute decompensated heart failure (ADHF).
* Patients deemed by the health care team to require hemodynamic monitoring with a pulmonary artery catheter and inotropic therapy. Patients receiving at least 3 doses of continued beta blocker therapy with carvedilol, metoprolol succinate, or metoprolol tartrate and patients receiving no beta blocker therapy or have missed at least 5 doses of beta-blocker therapy.

Exclusion Criteria:

* Concomitant treatment with other beta blockers, non-selective alpha blockers (e.g. terazosin, prazosin, doxazosin), non-dihydropyridine calcium antagonists, antiarrhythmic agents except for chronic stables doses of amiodarone, dofetilide or mexiletine.
* Use of inotropes or IV vasoactive agents within 7 days or at time of enrollment Patients with hemodynamically unstable arrhythmias (e.g., Systolic Blood Pressure (SBP) < 80, Heart Rate (HR) > 110), uncorrected primary valvular disease, or current mechanical support including left ventricular assist device (LVADs), Impella devices and balloon pumps
* Patients who have missed more than 1 dose of beta blocker within 72 hours of starting inotrope
* No subjects will be excluded based upon race, gender or ethnicity.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the General Cardiology and Heart Failure Services at the University of North Carolina Hospitals with acute decompensated heart failure, and who are deemed by the health care team to require pulmonary artery catheter placement and inotropic therapy with either dobutamine or milrinone by continuous infusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-12; Primary Completion 2017-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Fick Cardiac Index ( Fick CI) from baseline to maximum tolerated dose of inotrope therapy | baseline to maximum tolerated dose. (up to 6 hours)
  Dobutamine will be titrated every 2 hours as tolerated for a total of 3 titrations. Data will be collected over the 6 hour infusion.
  Milrinone titration timeframes are dependent on renal function and as tolerated by patients. A total of 3 titrations may occur as tolerated over incremental timeframes of 4, 12, 18 and 24 hours. Data will be collected over the 12-72 hours the patient will be receiving the milrinone infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Ellen Rodgers, PharmD, Principal Investigator — UNC Healthcare
Locations (1):
- UNC Healthcare, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Bollano E, Tang MS, Hjalmarson A, Waagstein F, Andersson B. Different responses to dobutamine in the presence of carvedilol or metoprolol in patients with chronic heart failure. Heart. 2003 Jun;89(6):621-4. doi: 10.1136/heart.89.6.621. PMID 12748215
- [Background] Metra M, Nodari S, D'Aloia A, Muneretto C, Robertson AD, Bristow MR, Dei Cas L. Beta-blocker therapy influences the hemodynamic response to inotropic agents in patients with heart failure: a randomized comparison of dobutamine and enoximone before and after chronic treatment with metoprolol or carvedilol. J Am Coll Cardiol. 2002 Oct 2;40(7):1248-58. doi: 10.1016/s0735-1097(02)02134-4. PMID 12383572
- [Background] Lowes BD, Tsvetkova T, Eichhorn EJ, Gilbert EM, Bristow MR. Milrinone versus dobutamine in heart failure subjects treated chronically with carvedilol. Int J Cardiol. 2001 Dec;81(2-3):141-9. doi: 10.1016/s0167-5273(01)00520-4. PMID 11744130
- [Background] Woolfrey SG, Hegbrant J, Thysell H, Fox PA, Lendrem DW, Lockwood GF, Lasher K, Rogers J, Greenslade D. Dose regimen adjustment for milrinone in congestive heart failure patients with moderate and severe renal failure. J Pharm Pharmacol. 1995 Aug;47(8):651-5. doi: 10.1111/j.2042-7158.1995.tb05853.x. PMID 8583366